CLINICAL TRIAL: NCT04909476
Title: Airways Management in COVID-19 Related Respiratory Failure: a Prospective Observational Multi-center Study
Brief Title: Tracheal Intubation in COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Bortolo Hospital (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Silvia De Rosa, Principal Investigator, St. Bortolo Hospital
Other Study IDs: 125/20
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: COVID-19 Pneumonia; Tracheal Intubation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe COVID pneumonia with ET: Severe COVID 19 pneumonia undergoing endotracheal intubation
  Interventions: Procedure: Endotracheal intubation

INTERVENTIONS:
Procedure: Endotracheal intubation — Airways management in COVID 19 patients pneumonia

SUMMARY:
The Emergency Endotracheal intubation of a patient who is COVID-19 positive is a high-risk procedure and an additional challenge to an intensivist due to barrier enclosures that have been developed to reduce the risk of COVID-19 transmission to healthcare providers during intubation. Although the incidence of difficult airways is commonly higher in critically ill patients, the evidence of severe hypoxemia without sign of respiratory distress could complicate the scenario.This silent hypoxia often leads to a delayed recognition of the severity of respiratory failure and to a late intubation which is often characterized by a high risk of complications related to the actual airways' management, hemodynamic and cardiac. It has been shown that non-survivors had worse blood gas analyzes than survivors, both before and after intubation. Few studies have reported the implications and adverse events of performing endotracheal intubation for critically ill COVID-19 patients admitted to intensive care units (ICUs).

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patient above 18 year old, admitted in the Intensive Care of San Bortolo Hospital, Vicenza, and San Matteo Hospital, Pavia;
* positive specimen for SARS-COV2 PCR;
* tracheal intubation for respiratory distress related to SARS COV2 pneumonia

Exclusion Criteria:

* negative specimen for SARS-COV2 PCR
* out of hospital intubation
* intubation during cardiac arrest
* intubation in the contest of general anesthesia for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patient above 18 year old, admitted in the Intensive Care
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-06-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse peri-intubation events | intubation procedure, an expected average 30 minutes
  The incidence of major adverse peri-intubation events defined as least one events:
  * cardiovascular instability
  * severe Hypoxemia
  * cardiac arrest

SECONDARY OUTCOMES:
Number of minor complications in the intubation process in patients admitted in the intensive care | 28 days
  This study will analyze the prevalence of minor complications related to intubation technique in the the Critical Unit. This information will be useful in order to determinate the risk factors associated.
Correlation between videolaryngoscope use and incidence of complication compared to the conventional laryngoscopy | 28 days
  Although the video laryngoscope is useful to perform difficult airways management, the benefits associated to its employment is still controversial compared to the conventional laringoscope.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Cattin, MD, Principal Investigator — SBortolo Hospital; Silvia De Rosa, MD, Principal Investigator — SBortolo Hospital; Silvia Mongodi, MD, Principal Investigator — SMatteo Hospital
Locations (2):
- Italy (2):
  - San Matteo Hospital, Pavia, Lombardy
  - San Bortolo Hospital, Vicenza, Veneto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yao W, Wang T, Jiang B, Gao F, Wang L, Zheng H, Xiao W, Yao S, Mei W, Chen X, Luo A, Sun L, Cook T, Behringer E, Huitink JM, Wong DT, Lane-Fall M, McNarry AF, McGuire B, Higgs A, Shah A, Patel A, Zuo M, Ma W, Xue Z, Zhang LM, Li W, Wang Y, Hagberg C, O'Sullivan EP, Fleisher LA, Wei H; collaborators. Emergency tracheal intubation in 202 patients with COVID-19 in Wuhan, China: lessons learnt and international expert recommendations. Br J Anaesth. 2020 Jul;125(1):e28-e37. doi: 10.1016/j.bja.2020.03.026. Epub 2020 Apr 10. PMID 32312571
- [Background] Carrillo A, Gonzalez-Diaz G, Ferrer M, Martinez-Quintana ME, Lopez-Martinez A, Llamas N, Alcazar M, Torres A. Non-invasive ventilation in community-acquired pneumonia and severe acute respiratory failure. Intensive Care Med. 2012 Mar;38(3):458-66. doi: 10.1007/s00134-012-2475-6. Epub 2012 Feb 9. PMID 22318634
- [Background] Huang HB, Peng JM, Weng L, Liu GY, Du B. High-flow oxygen therapy in immunocompromised patients with acute respiratory failure: A review and meta-analysis. J Crit Care. 2018 Feb;43:300-305. doi: 10.1016/j.jcrc.2017.09.176. Epub 2017 Sep 22. PMID 28968525
- [Background] Goh KJ, Choong MC, Cheong EH, Kalimuddin S, Duu Wen S, Phua GC, Chan KS, Haja Mohideen S. Rapid Progression to Acute Respiratory Distress Syndrome: Review of Current Understanding of Critical Illness from Coronavirus Disease 2019 (COVID-19) Infection. Ann Acad Med Singap. 2020 Mar 16;49(3):108-118. PMID 32200400
- [Background] Martin LD, Mhyre JM, Shanks AM, Tremper KK, Kheterpal S. 3,423 emergency tracheal intubations at a university hospital: airway outcomes and complications. Anesthesiology. 2011 Jan;114(1):42-8. doi: 10.1097/ALN.0b013e318201c415. PMID 21150574
- [Derived] Cattin L, Ferrari F, Mongodi S, Pariani E, Bettini G, Daverio F, Donadello K, Polati E, Mojoli F, Danzi V, De Rosa S. Airways management in SARS-COV-2 acute respiratory failure: A prospective observational multi-center study. Med Intensiva. 2023 Mar;47(3):131-139. doi: 10.1016/j.medin.2022.07.002. Epub 2023 Feb 24. PMID 36855737
- [Derived] Cattin L, Ferrari F, Mongodi S, Pariani E, Bettini G, Daverio F, Donadello K, Polati E, Mojoli F, Danzi V, De Rosa S. Airways management in SARS-COV-2 acute respiratory failure: A prospective observational multi-center study. Med Intensiva (Engl Ed). 2023 Mar;47(3):131-139. doi: 10.1016/j.medine.2022.08.005. Epub 2022 Aug 8. PMID 36155747